CLINICAL TRIAL: NCT01751048
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the Vaccine Candidates LEISH-F3 + GLA-SE, LEISH-F3 + MPL-SE, and LEISH-F3 + SE in Healthy Adult Subjects
Brief Title: LEISH-F3 + GLA-SE and the LEISH-F3 + MPL-SE Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0031; HHSN272200800008C
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2015-05

CONDITIONS: Leishmaniasis
Keywords: GLA-SE,LEISH-F3,leishmaniasis,MPL-SE,parent protocol,vaccine
MeSH Terms: conditions — Leishmaniasis | interventions — glucopyranosyl lipid-A

ARMS (3):
- Group #1 (Experimental): N=16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg of LEISH-F3 + 5 mcg Glucopyranosyl Lipid A- Stable oil-in-water emulsion (GLA-SE)
  Interventions: Biological: GLA-SE; Biological: LEISH-F3
- Group #2 (Experimental): N=16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg of LEISH-F3 + 10 mcg Monophosphoryl Lipid A-Stable oil-in-water emulsion (MPL-SE)
  Interventions: Biological: LEISH-F3; Biological: MPL-SE
- Group #3 (Experimental): N=16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg LEISH-F3 + Stable oil-in-water Emulsion (SE)
  Interventions: Biological: LEISH-F3; Drug: SE

INTERVENTIONS:
Biological: GLA-SE — Glucopyranosyl Lipid A- Stable oil-in-water emulsion (GLA-SE) is formulated in a stable oil-in-water emulsion (SE) to yield the adjuvant formulation GLA-SE. The combination of GLA-SE with a recombinant protein antigen (LEISH-F3) results in a Th1-type T cell response. GLA-SE appears as a milky- white liquid. 16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg of LEISH-F3 + 5 mcg GLA-SE.
  Arms: Group #1
Biological: LEISH-F3 — LEISH-F3 is a lyophilized formulation containing 50 mcg LEISH-F3 and excipients (mannitol, sucrose, and polysorbate 80). All subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg of LEISH-F3.
Biological: MPL-SE — Monophosphoryl Lipid A-Stable oil-in-water emulsion (MPL-SE) is an oil-in-water emulsion that contains Monophosphoryl Lipid A, an attenuated form of Lipid A from Salmonella Minnesota R595 in a emulsion (SE). The combination of MPL-SE with a recombinant protein antigen (LEISH-F3) results in a TH1-type T cell response. MPL-SE appears as a milky-white liquid. 16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg of LEISH-F3+10 mcg MPL-SE.
  Arms: Group #2
Drug: SE — Stable oil-in-water Emulsion (SE) is a squalene oil-in-water emulsion that has adjuvant properties of its own, but in a Th2-dependent manner. SE appears as milky-white liquid. 16 subjects receive vaccine on day 0, 28, and 168 of 0.5 ml of 20 mcg LEISH-F3 + SE.
  Arms: Group #3

SUMMARY:
Investigational products: LEISH-F3 (recombinant protein antigen) + GLA-SE (adjuvant) leishmaniasis vaccine and LEISH-F3 (recombinant protein antigen) + MPL-SE (adjuvant) leishmaniasis vaccine. Stage of development: Phase 1 clinical development. Healthy adult subjects, 18 to 49 will be recruited through a U.S. site. Primary objective: To evaluate the safety and tolerability of the LEISH-F3 + GLA-SE vaccine and the LEISH-F3 + MPL-SE vaccine following intramuscular (IM) administration of 20 µg of LEISH-F3 together with 2 or 5 µg of GLA-SE or 10 µg of MPL-SE on Days 0, 28, and 168. Secondary objective: To assess the immunogenicity of LEISH-F3 formulated with GLA-SE, MPL-SE, or SE by evaluating IgG antibody responses to LEISH-F3 at Days 0, 28, 56, 168, 196, and 365, and T cell responses to LEISH-F3 at Days 0, 14, 42, 168, 182, and 365. Each subject's duration of participation will be about 18 months.

DETAILED DESCRIPTION:
Leishmaniasis is a disease caused by protozoan parasites of the genus Leishmania. The parasites are transmitted from an animal or human reservoir through the bite of infected female phlebotomine sand flies. This study is a randomized, open-label clinical trial designed to evaluate the safety, tolerability, and immunogenicity of the LEISH-F3 recombinant protein antigen formulated with GLA-SE, MPL-SE, or SE adjuvant in healthy adults 18 to 49 years of age. Each subject's duration of participation will be about 18 months. Subjects will receive a total of 3 doses of vaccine, which will be given by intramuscular injection on Days 0, 28, and 168. The volume of each vaccine dose will be 0.5 mL. A computerized system will be used to acquire any data regarding halting criteria throughout the study. Primary objective is to evaluate the safety and tolerability of LEISH-F3 formulated with GLA-SE, MPL-SE, or SE following intramuscular administration of 20 µg of LEISH-F3 together with 5 µg of GLA-SE, 10 µg of MPL-SE, or SE alone. Secondary objective is to assess the immunogenicity of LEISH-F3 formulated with GLA-SE, MPL-SE, or SE by evaluating IgG antibody responses to LEISH-F3 at Days 0, 28, 56, 168, 196, and 365, and T cell responses to LEISH-F3 at Days 0, 14, 42, 168, 182, and 365. A substudy will be performed using up to 12 subjects from each Study Group (Groups 1, 2 and 3) and an additional 12 subjects to serve as controls. This substudy will investigate whether, as in murine cells, cell surface markers (CD11a, CD49d) can be used as a surrogate to identify protective immune CD4+ T cells in human subjects receiving a vaccine antigen.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females between the ages of 18 and 49 years, inclusive. 2. Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who have not been postmenopausal for >/=1 year) must agree to practice adequate contraception for the 28-day period before vaccination through 90 days after the third vaccination. Acceptable birth control methods for the purposes of this study may include, but are not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, and intrauterine devices, and licensed hormonal methods. 3. In good health, as judged by the investigator and determined by vital signs [temperature < 38 degrees Celsius, heart rate </= 100 bpm and > 50 bpm, systolic blood pressure </= 140 mmHg and > 89 mmHg, diastolic blood pressure </= 90 mmHg and >/= 60 mm Hg, medical history and a targeted physical examination. Athletically trained subjects with a pulse >/= 45 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator]. 4. Screening laboratory values must be within normal limits. These include blood hemoglobin, white blood cell (WBC) count, neutrophil count, platelets, creatinine, AST (Aspartate Aminotransferase), ALT (Alanine Aminotransferase), bilirubin (total), glucose (random, must be less than 140), and urine dipstick for protein and glucose. Note: trace proteinuria is acceptable; creatinine, AST, ALT, and bilirubin values lower than the normal range are acceptable. The following serology tests must be negative: HIV (Human immunodeficiency virus) ( 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. HIV and hepatitis C viral load PCR (Polymerase chain reaction) testing may be performed for individuals suspected of having indeterminate antibody testing. 5. Able to understand and comply with planned study procedures. 6. Willing to be available for all study-required procedures, visits and calls for the duration of the study. 7. Provide written informed consent before initiation of any study procedures and be available for all study visits. 8. Willing to abstain from donating whole blood or blood derivatives until 90 days after the final study vaccination. Eligibility Criteria for Doses 2 and 3 Subjects must meet all inclusion and exclusion criteria as outlined in sections 5.1 and 5.2 with the exception of clinical safety lab values. Subjects with safety laboratory values that meet Grade 2 or greater severity (according to the toxicity table, Appendix C), that do not return to the protocol-defined normal range prior to the second or third vaccination will not be eligible to receive additional doses of study vaccine. Repeat HIV, hepatitis B and hepatitis C serologies are not required prior to the second and third vaccinations. Eligibility for Unvaccinated Substudy Control Population 1. Males and females between the ages of 18 and 49 years, inclusive. 2. In good health, as judged by the investigator and determined by vital signs [temperature < 38degrees C, heart rate </= 100 bpm and > 50 bpm, systolic blood pressure </= 140 mmHg and > 89 mmHg, diastolic blood pressure </= 90 mmHg and >/= 60 mm Hg, medical history and a targeted physical examination. Athletically trained subjects with a pulse >/= 45 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator. 3. Has received tetanus toxoid vaccination within the past 10 years. 4. Able to understand and comply with planned study procedures. 5. Willing to be available for a ll study-required procedures, visits and calls for the duration of the study. 6. Provide written informed consent before initiation of any study procedures and be available for all study visits.

Exclusion Criteria:

1. History of possible infection with Leishmania or previous exposure to Leishmania vaccines or experimental products containing GLA-SE. 2. Veterans who served in the military in the Middle East (Iran, Iraq), Afghanistan, or any other areas endemic to Leishmania. 3. Travelers to, or immigrants from, areas endemic to Leishmania (Appendix D). Certain countries have endemic leishmaniasis only in certain regions of the country.The study PI (Principle Investigator) or a designated clinician may review the travel history with a potential candidate to determine if travel included areas of the country with endemic leishmaniasis. 4. Body temperature >/= 100.4 degrees Farenheit (>/=38.0 degrees Celsius) or acute illness within 3 days before vaccination (subject may be rescheduled). 5. A positive serum or urine pregnancy test within 24 hours prior to vaccination (if female of childbearing potential as defined in Inclusion Criterion 2), women who are planning to become pregnant from 30 days prior to entering the study until 90 days after the final study vaccination, or women who are breastfeeding. 6. Immunosuppression as a result of an underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months. 7. An active neoplastic disease (excluding nonmelanoma skin cancer) or a history of any hematologic malignancy. Active neoplastic disease is defined as neoplastic disease or treatment for neoplastic disease within the past 5 years 8. A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarteritis, thyroiditis, etc). 9, Used an immunosuppressive or immunomodulatory drug such as >0.5 mg/kg/day or >/= 20 mg total dose/day of prednisone orally or >800 microgram of inhaled beclomethasone for 2 or more consecutive weeks within 6 months prior to the first vaccination (Nasal and topical steroids are allowed). 10. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt. 11. A history of treatment for any other psychiatric disorder in the past 3 years that increases the risk to the subject in the opinion of the investigator. 12. A history of receiving immunoglobulin or other blood product within the previous 3 months before vaccination or a history of donating whole blood within the past two months or other blood derivatives within 2 weeks. 13. Received or plan to receive any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks of any study vaccination. 14. An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses or is not generally seen in healthy, normal subjects. (This includes, but is not limited to, known cardiac disease, pulmonary disease, liver disease, renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.) 15. Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines, eggs, or unknown allergens or known allergy to components of the vaccine. 16. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month before vaccination in this study or expect to receive an experimental agent during the 18 month study period. 17. Any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or that may interfere with successful completion of the study. 18. A history of alcohol or drug abuse du ring the previous 1 year, for example, daily excessive alcohol use or frequent binge drinking as determined by the investigator, or chronic marijuana abuse or any other illicit drug use. 19. Presence of tattoos that would preclude evaluation of the injection site. Subject Exclusion Criteria for Unvaccinated Substudy Control Population 1. History of possible infection with Leishmania or previous exposure to Leishmania vaccines. 2. Veterans who served in the military in the Middle East (Iran, Iraq), Afghanistan, or any other areas endemic to Leishmania. 3. Travelers to, or immigrants from, areas endemic to Leishmania (Appendix D). Certain countries have endemic leishmaniasis only in certain regions of the country. The study PI or a designated clinician may review the travel history with a potential candidate to determine if travel included areas of the country with endemic leishmaniasis. 4. Body temperature >/=100.4 degrees F (>/=38.0 degrees C) or acute illness within 3 days before vaccination (subject may be rescheduled). 5. Immunosuppression as a result of an underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months. 6. An active neoplastic disease (excluding nonmelanoma skin cancer) or a history of any hematologic malignancy. Active neoplastic disease is defined as neoplastic disease or treatment for neoplastic disease within the past 5 years. 7. A history of autoimmune disease (systemic lupus, rheumatoid arthritis, scleroderma, polyarteritis, thyroiditis, etc). 8. Used an immunosuppressive or immunomodulatory drug such as >0.5 mg/kg/day or >/=20 mg total dose/day of prednisone orally or >800 mcg of inhaled beclomethasone for 2 or more consecutive weeks within 6 months prior to phlebotomy (Nasal and topical steroids are allowed). 9. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt. 10. A history of treatment for any other psychiatric disorder in the past 3 years. 11. A history of receiving immunoglobulin or other blood product within the previous 3 months before vaccination or a history of donating whole blood within the past two months or other blood derivatives within 2 weeks. 12. Received or plan to receive any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks of any study vaccination. 13. An acute or chronic medical condition that, in the opinion of the investigator, would interfere with the evaluation of responses or is not generally seen in healthy, normal subjects. (This includes, but is not limited to, known cardiac disease, pulmonary disease, liver disease, renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse events considered related to the vaccination at any point during the study period. | approximately 533 days
The number of subjects experiencing solicited injection site reaction within 7 days following vaccination. | Through 7 days following vaccination
The number of subjects experiencing solicited systemic reactions within 7 days following vaccination. | Through 7 days following vaccination
The number of subjects spontaneously reporting adverse events considered related to the vaccination at any point during the study period. | Through Day 365

SECONDARY OUTCOMES:
The magnitude of Th1 and Th2 cytokine production in PBMCs in response to the LEISH-F3 antigen relative to baseline as assayed by Luminex. | Days 14, 42, 168, 182, and 365
The proportion of subjects with at least a 4-fold increase in IgG antibody responses to LEISH-F3 relative to baseline. | Days 28, 56, 168, 196, and 365

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa, United States